CLINICAL TRIAL: NCT04723303
Title: Phase 1 Study of Mesenchymal Stromal Cells, Umbilical Cord Lining Stem Cells (ULSC), in Patients With Polymyositis (PM) and Dermatomyositis (DM)
Brief Title: Phase 1 Study of ULSC in Patients With Polymyositis (PM) and Dermatomyositis (DM)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Restem, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DM/PM V2.0; IRB201903442 (Other: UF IRB); OCR33722 (Other: UF OnCore)
Record Dates: First submitted 2020-12-08; First posted 2021-01-25 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Polymyositis; Dermatomyositis
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Intervention Model Description: Study Participants will be assigned to one of 3 doses of stem cells depending on when the subject is enrolled. The first three patients will be assigned to the low dose group, the next three patients will be assigned the intermediate dose group and last three patients will receive the high dose of ULSC's. An independent review group will evaluate the response to therapy to each dose group before moving to the next dose. The groups and doses are described below:
  A low dose group receives an IV infusion of 50 million stem cells.
  An intermediate dose group receives an IV infusion of 100 million stem cells.
  A high dose group receives an IV infusion of 200 million stem cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): A single IV infusion of ULSC's in patients with DM or PM
  Interventions: Drug: Umbilical Cord Lining Stem Cells

INTERVENTIONS:
Drug: Umbilical Cord Lining Stem Cells — An IV infusion of ULSCs will be administered.

SUMMARY:
This study will investigate Umbilical Cord Lining Stem Cells (ULSC) as an investigational medicinal product and its use in patients with polymyositis (PM) or dermatomyositis (DM) to see if a single intravenous (IV) infusion of allogeneic umbilical cord lining stem cells (ULSC) safe, tolerable, and feasible to administer.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male or female, age ≥18 years old
2. Diagnosis of definite or probable DM or PM, according to the criteria of Bohan and Peter
3. Patients with PM will either be positive for a myositis-associated antibody or have undergone evaluation to exclude mimics, as deemed appropriate by the Investigator (See Note below).
4. Signs informed consent.

Exclusion Criteria:

1. A diagnosis of inclusion body myositis, juvenile DM or PM, myositis in the context of significant overlap with another systemic autoimmune rheumatologic disease.
2. Non immune myopathies.
3. Cancer associated myositis.
4. Hypersensitivity to study product components. History of hypersensitivity to dimethyl sulfoxide (DMSO).
5. Pregnant or lactating women.
6. Concomitant severe cardiac, pulmonary disease, active infection or other conditions that preclude assessment of safety and efficacy of the study product.
7. Patients with predominant muscle atrophy secondary to uncontrolled or chronic DM or PM, based on clinical, biochemical, and/or radiologic assessment, despite previous optimized treatment.
8. Anticipated need for surgery during the trial period.
9. A history of prevalent noncompliance with medical therapy.
10. Recipient of an organ transplant.
11. Neutropenia (absolute neutrophil count<1,800/mm3 [or <1,000/mm3 in African-American subjects]).
12. Severe impairment in renal function (estimated glomerular filtration rate <30 ml/kg*min).
13. Recent or planned use of vaccination with live attenuated viruses.
14. Active cancer or prior diagnosis of cancer within the past 2 years (patients with basal and squamous cell cancer of skin will not be excluded).
15. Condition that would impair an assessment of muscle strength, including neurological disorders such as Parkinson's disease or severe musculoskeletal condition.
16. Any other condition that, in the judgment of the Investigator or Sponsor, would be a contraindication to enrollment, study product administration, or follow-up.
17. History of Atrial septal defect or ventricular septal defect

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Dose Limiting Toxicity (DLT) that begins during or following ULSC infusion as assessed within 24 hours. | Within 24 hours
  Dose Limiting Toxicities are treatment-emergent suspected adverse reactions graded severe, such as severe infusion-related hypersensitivity toxicities of grade ≥3, and any serious adverse event (SAE). (Note: DLT during an infusion will stop that infusion in that subject.)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No